CLINICAL TRIAL: NCT05423210
Title: A Pilot Study to Evaluate the Immunogenic Effects of Window-of-Opportunity Fractionated Stereotactic Radiotherapy Combined With Atezolizumab for Patients With Newly Diagnosed WHO CNS Grade 4 Glioma (Glioblastoma Multiforme)
Brief Title: Atezolizumab and Pre-Surgical Brain Radiation Therapy for Glioblastoma Multiforme
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Alexander Stessin, Professor of Medicine, Stony Brook University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBU-FSRT-NEURO
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Combination Product: Atezolizumab + FSRT radiation

INTERVENTIONS:
Combination Product: Atezolizumab + FSRT radiation — Atezolizumab 840mg IV every 2 weeks Fractionated Stereotactic Radiotherapy

SUMMARY:
This is a single-arm pilot study that will recruit 12 patients with newly diagnosed Glioblastoma, a malignant brain tumor with a poor prognosis. Patients will be treated with fractionated stereotactic radiotherapy (FSRT) for 2 weeks, in addition to two doses of Atezolizumab (Tecentriq), an FDA approved PD- L1 inhibitor drug, 840 mg IV, at the beginning and at the end of the two-week time period, concomitantly with FSRT. After this initial two weeks treatment the patients will undergo craniotomy and maximal safe resection as per normal care for a GB. After surgery patients will follow the normal care for glioblastoma in addition to Atezolizumab 840 mg IV q2 weeks for the duration of adjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of glioblastoma multiforme WHO Grade IV
* The patient is a surgical candidate, with the surgical intent for a > 80% resection of the lesion
* Negative pregnancy test
* ECOG status <= 2
* Tumor volume <= 3.5 cm
* Adequate organ function
* Negative for infectious disease (human immunodeficiency virus, Hepatitis B Virus, Hepatitis C Virus, tubercolosis)

Exclusion Criteria:

* Patient already underwent surgical total or partial tumor resection, or radiation therapy
* Presence of leptomeningeal disease, gliomatosis cerebri, multifocal disease, bilateral cerebral hemisphere involvement ("butterfly" gliomas)
* Patients at increased risk of neurologic decompensation
* Continued use of high dose intravenous or oral corticosteroids, or > 8milligrams per day of systemic dexamethasone
* Uncontrolled tumor-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)
* Uncontrolled or symptomatic hypercalcemia
* History of autoimmune disease or immune deficiency
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis
* Significant cardiovascular disease
* History of other malignancy within 1 year prior to screening
* Severe infection within 4 weeks prior to initiation of study treatment
* History of allogeneic stem cell or organ transplant
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies
* Treatment with systemic immunostimulatory agents
* Treatment with systemic immunosuppressive medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants who progress/relapse after surgical resection | 2 years
  Assess the efficacy of atezolizumab in combination with fractionated stereotactic radiation therapy in the neoadjuvant setting for resectable glioblastoma multiforme
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 30 days after the last dose of atezolizumab
  Assess the safety of atezolizumab in combination with fractionated stereotactic radiation therapy in the neoadjuvant setting for resectable glioblastoma multiforme

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Stessin, MD, Principal Investigator — Stony Brook Cancer Center
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No